CLINICAL TRIAL: NCT03392012
Title: Effect of Sedation on Pulmonary Aeration in Children
Acronym: LunSed
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Gemma, Principal Investigator, IRCCS San Raffaele
Other Study IDs: 140/INT/2017
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Sedative Adverse Reaction
Keywords: anesthesia, patient safety, respiratory complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pediatric sedation is an anesthesiological technique with a good safety profile, but various complications might ensure, especially from the respiratory point of view. No suggestion is available about a possible upper safety limit for the duration of sedation to limit respiratory issue. In order to address this topic, the investigators concentrated on the occurrence of hypoventilated lung areas, which is a well-known side effect of anesthesia and sedation. The investigators hypothesis that the length of sedation is correlated with the occurrence of lung atelectasis and hypoventilation. To assess lung hypoventilation the lung ultrasound will be used. Lung ultrasound will be performed immediately after the induction of sedation and immediately before sedation interruption, in children scheduled for magnetic resonance exams.

The study is a prospective observational study

DETAILED DESCRIPTION:
Worldwide, an increasing number of medical procedures are performer in children under sedation in many different clinical settings, in compromised patients, often outside the operating theater and often by non-anesthesiologists.

Although a good safety profile accounts for the spread of sedation, various complications might ensure. Furthermore of all the patients receiving sedation for diagnostic and therapeutic procedures, the pediatric population is the subgroup at the highest risk level and with the lowest tolerance of error.

In the last years the results of two large database studies have been published to lend some clarity on the rate and nature of adverse events involving sedation/anesthesia outside the operating room. Respiratory complications were the most frequently reported, and required critical anesthesiological competencies for a correct management to avoid poor outcomes.

Risk factors for adverse events during sedation/anesthesia have been evaluated by the 2016 SIAARTI(Società Italiana di Anestesia, Analgesia, Rianimazione e Terapia Intensiva)-SARNePI (Società di Anestesia e Rianimazione Neonatale e Pediatrica Italiana) guidelines for the standard of pediatric anesthesia, including patients' age, ASA (American Society of Anesthesiology) class, experience of the operators, and urgency/emergency conditions.

On the other hand, no suggestion is available either in current literature or guidelines, about a possible upper safety limit for the duration of sedation. In order to address this topic, the investigators concentrated on the occurrence of hypoventilated lung areas, which is a well-known side effect of anesthesia and sedation. To assess lung hypoventilation the LUSS-Lung Ultrasound Score will be used, since it is a validated and non invasive tool.

The study aims to assess the incidence of atelectasis and hypoventilated lung areas after sedation in children and evaluating possible risk factors for them. The investigators hypothesis that the length of sedation is correlated with the occurrence of lung atelectasis and hypoventilation.

This prospective observational cohort study study could suggest an upper safety limit for the duration of pediatric sedations, which is not reported in the available literature.

Consecutive children (age 1-8 yrs old) scheduled to undergo cerebral or medullary magnetic resonance imaging under deep sedation will be enrolled. In the investigators' center such MR imaging data acquisition (and the relevant sedation) ranges usually between 40 and 120 minutes. Enrollment will take place on the day of sedation.

Informed consent will be obtained from both parents at the preoperative visit or the day of the procedure.

The children will be sedated with propofol iv according to a standard clinical protocol and spontaneous breathing will be maintained throughout the study. The standard protocol has been internally validated both in the clinical and scientific setting.

Immediately after the induction of sedation, lung ultrasound will be performed and the imaging will be scored according to the lung ultrasound score(LUSS). Thereafter the child will be transferred into the magnetic resonance (MR) suite and the MR exam will be performed as required. After completion of MR imaging child will be transferred back to the recovery room and the sonographer will re- assess the LUSS before the discontinuation of sedation. Hence, two lung ultrasound evaluations will be performed: one at the beginning and one at the end of sedation.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-8 years old (included)
* Informed consent of both parents
* Scheduled for elective cerebral or medullary Magnetic Resonance exam

Exclusion Criteria:

* Any ongoing respiratory disease
* Contraindications to the use of propofol
* LUSS ≤12 at the first US assessment (a baseline maximum score 1 on all of the pulmonary fields)
* need for mechanical ventilation

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children scheduled to undergo cerebral or medullary magnetic resonance imaging under deep sedation
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Lung Ultrasound Score in children undergoing deep sedation | through study completion, an average of 1 hour
  Lung ultrasound score

SECONDARY OUTCOMES:
Effect of sedation length on hypoventilation in children undergoing deep sedation | through study completion, an average of 1 hour
  Sedation length (min)
Incidence of any respiratory and non-respiratory adverse event in children undergoing deep sedation | through study completion, an average of 1 hour
  Clinical observation

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gemma, MD, Study Chair — IRCCS San Raffaele, Milan, Italy
Locations (1):
- S. Raffaele Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No